CLINICAL TRIAL: NCT03105297
Title: An Exploratory Study of a Nasal Dilator Strip
Brief Title: To Characterize the Performance of the Nasal Dilator Strip in Lowering Nasal Resistance During Sleep, Promoting Nasal Route Breathing and Reducing the Signs and Symptoms of Sleep Disordered Breathing in a Group of Chronic Nocturnal Nasal Congestion Sufferers Who Report Trouble With Their Sleep.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202203; NCT01004471 (obsolete NCT alias)
Record Dates: First submitted 2017-04-05; First posted 2017-04-07 (Actual); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Sleep Disordered Breathing; Congestion, Nasal
Keywords: Nasal dilator strip; Sleep disordered breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: This study consisted of 3 phases baseline and active phase in which participants used the nasal dilator strip followed by 2 nights cross over nasal resistance phase in which participants were randomized to receive a sequence of strip/no strip or no strip/strip.
Oversight: Data Monitoring Committee: No

ARMS (3):
- All participants (Baseline phase) (Experimental): All the participants were applied nasal dilator strip during the sleep laboratory night on Day 1.
  Interventions: Device: Prototype nasal dilator strip
- All Participants (Active Phase) (Experimental): All the participants wore nasal dilator strip over a 1 month in-home use period and returned for sleep laboratory nights after 7 (Day 8) and 28 days (Day 29) of treatment
  Interventions: Device: Prototype nasal dilator strip
- All Participants (Nasal Resistance Phase) (Experimental): The participants were randomized to receive a sequence of either 'strip'/' no strip' or 'no strip'/'strip' on 2 sleep laboratory nights (on Day 30 and Day 31) based on the randomization schedule
  Interventions: Device: Prototype nasal dilator strip; Other: No strip

INTERVENTIONS:
Device: Prototype nasal dilator strip — External Prototype Nasal Dilator strip. GSK prototype nasal dilator AB 2R11. All the participants used nasal dilator strip throughout the active phase of the study (Day 1 to Day 28). Followed by that all the participants used the nasal strip on Day 29 or 30 in Nasal resistance phase of the study as per their randomization sequence.
Other: No strip
  Arms: All Participants (Nasal Resistance Phase)

SUMMARY:
To characterize the performance of the nasal dilator strip in lowering nasal resistance during sleep, promoting nasal route breathing and reducing the signs and symptoms of sleep disordered breathing in a group of chronic nocturnal nasal congestion sufferers who report trouble with their sleep.

DETAILED DESCRIPTION:
This study was a baseline-controlled study. This study consisted of three phases: Baseline phase, 28 days Active phase (1 month in home treatment usage period with sleep laboratory nights after 7 (Night 8) and 28 days (Night 29) of treatment) followed by a two-night cross-over Nasal resistance phase. Screened participants were evaluated for sleep disordered breathing and PSG variables with sleep laboratory nights at Baseline, after 7 and 28 days of in house use of nasal dilator strip (Night 8 and 29 of Active phase), and at Day 30 and 31 (Night 30 and 31 of Nasal resistance phase). Participants wore the Nasal dilator strip during Active phase. Participants then entered the Nasal resistance phase of the study, which consisted of two sleep laboratory nights at Day 30 and 31 (Night 30 and 31) where they were randomized to receive a sequence of either 'strip'/' no strip' or 'no strip'/'strip" as per there randomization schedule.

ELIGIBILITY:
Inclusion Criteria:

* Nostril types I and II (Inter-axial angle below 41 degrees = type I; inter-axial angle from 41 to 70 degrees = type II)
* Nasal Congestion: Have chronic nocturnal nasal congestion ('always or almost always') for at least the last year.
* Sleep: Reports trouble with sleep

Exclusion Criteria:

* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to latex. Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds), allergy or atopic reaction to adhesive bandages or latex.
* Subject has a chronic skin condition or eczema on the face or nose.
* Subject has visible open sores, sunburn, irritation on the face or nose immediately prior to treatment.
* Subject has severe obstructive sleep apnea/hypopnea syndrome with an AHI score <30 events/hour at the Baseline visit.
* Subject has had a diagnosis of another major sleep disorder (i.e. primary insomnia, i.e. regularly sleeping less than 6 hours per night, sleep insufficiency, i.e. sleeping >2 hours more on non-work days as compared to work days, narcolepsy, or periodic limb movement disorder).
* Subject has a non-typical sleep schedule (e.g. shift-work).
* Subject plans travel involving time-zone changes during the study period.
* Subject takes medication known to have a significant effect on sleep. Use of any substance with psychotropic effects or properties known to affect sleep/wake, including but not limited to: neuroleptics, morphine/opioid derivatives, sedative antihistamines, stimulants, antidepressants, clonidine, barbiturates, anxiolytics, thalidomide, hypnotics and sedatives. Use of over the counter sleep promoting agents including diphenhydramine, doxylamine, tryptophan, valerian root, kava kava, melatonin, St John's Wort and Alluna. Use of over the counter alertness aids including caffeine and guarana.
* Subject currently uses any topical nasal decongestants (nasal sprays, drops, etc). Subject must have discontinued use of topical decongestants at least 7 days prior Baseline.
* Subject is experiencing an acute upper respiratory tract infection at during qualification phase and at Baseline visit.
* Subject abuses alcohol (regularly drinks more than 3 drinks per day) or has a recent history (within last 2 years) of substance or alcohol abuse. Regular consumption of xanthine-containing beverages (i.e. tea, coffee, or cola) comprising usually more than 5 cups or glasses per day.
* Subject has a positive drug of abuse screening result.
* Subject has severe, unstable disease states (e.g. myocardial infarction, congestive heart failure, diabetes, cirrhosis, cancer, epilepsy, or stroke), pain syndromes, (e.g. fibromyalgia) or any medical or surgical condition that places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study or who in the judgement of the principal investigator would not be suitable for entry into this study.
* Severe nasal obstruction caused by structural abnormality that renders the subject unsuitable for the study in the opinion of the investigator, i.e. nasal polyps, severe deviated septum.
* Subject is unwilling to be videotaped or recorded during the PSG studies.
* Current Treatment for Sleep Disordered Breathing a) Subject currently uses devices prescribed for sleep disordered breathing including Continuous Positive Airway Pressure (CPAP), mandibular advancement devices, tongue displacement devices. b)Over-the-counter products such as chin straps, pillows, internal/external nasal dilators are acceptable provided usage is discontinued at least 28 days prior to Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-09-25 (Actual); Primary Completion 2010-08-10 (Actual); Study Completion 2010-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Wheatley JR, Amis TC, Lee SA, Ciesla R, Shanga G. Objective and Subjective Effects of a Prototype Nasal Dilator Strip on Sleep in Subjects with Chronic Nocturnal Nasal Congestion. Adv Ther. 2019 Jul;36(7):1657-1671. doi: 10.1007/s12325-019-00980-z. Epub 2019 May 22. PMID 31119695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in Australia.
Pre-assignment Details: 103 participants were screened, out of which 9 were screening failure, 3 did not want to participate. Remaining 91 participants were included in the safety population.
Groups:
- All Participants: The study consisted of 3 phases: baseline phase, 28 days active phase followed by a two-night cross-over nasal resistance phase. In the baseline phase all the participants applied nasal dilator strip during the sleep laboratory night on Day 1. During the active phase participants wore nasal dilator strip over a 1-month in-home use period and returned for sleep laboratory nights after 7 days (on Day 8) and 28 days (on Day 29) of treatment. The nasal resistance phase consisted of 2 sleep laboratory nights (Day 30 and 31), where the participants were randomized to receive a sequence of either 'strip'/' no strip' or no strip'/'strip' as per the randomization schedule
Period: Baseline Phase (Day 1)
Arm/Group | All Participants
Started | 91
Completed | 70
Not Completed | 21
Not completed — Other | 21
Period: Active Phase (Day 2-29)
Arm/Group | All Participants
Started | 70
Completed | 70
Not Completed | 0
Period: Nasal Resistance Phase (Day 30, 31)
Arm/Group | All Participants
Started | 56 (14 participants withdrew from the study after the completion of active phase)
Treated | 55
Completed | 48
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Population: Safety population N=91, All participants to whom the study treatment was dispensed were considered evaluable for the safety population.
Groups:
- All Participants: All participants to whom the study treatment was dispensed were considered evaluable for baseline characteristics
Arm/Group | All Participants
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.8 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 70
  Black | 2
  Asian | 9
  Hispanic | 1
  Other | 9

OUTCOME MEASURES:

1. Primary Outcome: Nasal Resistance in Sleeping State : Nasal Resistance Phase
Description: Nasal resistance of the participants with and without strip was measured in sleeping state using a nasal mask and a flow meter to obtain a trans-nasal pressure difference and nasal flow by continuous recording over the 2 nights [on Day 30 (Visit 5) and Day 31 (Visit 6), cumulatively], of the nasal resistance phase.
Time Frame: upto 2 days
Population: Per protocol population included all participants who fully complied with all study procedures and restrictions. Here, number of participants analyzed "N" signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable for the specified categories.
Measure: Mean (Standard Deviation); unit: Centimeter (cm) H2O/liter/sec
Arm/Group | All Participants (Nasal Resistance Phase)
Number analyzed (Participants) | 55
Centimeter (cm) H2O/liter/sec
  Without strip (Day 30 and 31): number analyzed (Participants) | 44
  Without strip (Day 30 and 31) | 2.658 (2.4469)
  With strip (Day 30 and 31): number analyzed (Participants) | 46
  With strip (Day 30 and 31) | 2.202 (2.5819)
Statistical Analysis 1: Comparison: All Participants (Nasal Resistance Phase); Test type: Superiority; p = 0.0147, ANCOVA — p-value for comparing between treatments (strip/no strip) were computed from mixed models with treatment & period as fixed effects, participants as random effects & time as repeated measures effect

2. Primary Outcome: Area at Minimum Cross Sectional Area 1 (MCA1) : Baseline Phase
Description: Minimum cross sectional area 1 (MCA1) in the first 3 cm of the nasal cavity behind the nostril (0-3 cm), considered to be the area of the nasal valve and the distance from the nares of this restriction. MCA 1 was measured with an Acoustic Rhinometer at Day 1 (baseline phase) before and after Nasal dilator strip application.
Time Frame: Day 1
Population: Safety population included all participants to whom the study treatment was dispensed. Here, "N" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | All Participants (Baseline Phase)
Number analyzed (Participants) | 70
cm^2
  Before strip application | 1.949 (0.8520)
  After strip application | 2.535 (0.8735)
Statistical Analysis 1: Comparison: All Participants (Baseline Phase); Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — p-values are from a one sample t-test using SAS UNIVARIATE on change from baseline

3. Primary Outcome: Volume at Minimum Cross-sectional Area 1 (MCA1) : Baseline Phase
Description: Volume of the first 3 cm of the nasal cavity behind the nostril (0-3 cm2). Volume at MCA1 was measured with an Acoustic Rhinometer at Day 1 before and after Nasal dilator strip application.
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | All Participants (Baseline Phase)
Number analyzed (Participants) | 70
cm^3
  Before strip application | 4.145 (1.2013)
  After strip application | 5.043 (1.4038)
Statistical Analysis 1: Comparison: All Participants (Baseline Phase); Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — p-values are from a one sample t-test using SAS UNIVARIATE on change from baseline

4. Primary Outcome: Nasal Resistance by Posterior Rhinomanometry : Baseline Phase
Description: Nasal resistance was measured on Day 1, by a modified method of posterior rhinomanometry in awake and seated position. Using posterior rhinomanometry, the transnasal pressure difference was measured between the nasopharynx and the external nares. The technique measures the difference in transnasal pressure that drives the flow of air through the nasal cavities.
Time Frame: Day 1
Population: Safety population included all participants to whom the study treatment was dispensed. Here, "N" signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable for the specified categories.
Measure: Mean (Standard Deviation); unit: cmH2O/liter/seconds
Arm/Group | All Participants (Baseline Phase)
Number analyzed (Participants) | 70
cmH2O/liter/seconds
  Before strip application: number analyzed (Participants) | 51
  Before strip application | 4.468 (4.7625)
  After strip application: number analyzed (Participants) | 50
  After strip application | 3.251 (4.1677)
Statistical Analysis 1: Comparison: All Participants (Baseline Phase); Test type: Superiority or Other; p = 0.0073, t-test, 1 sided — p-values are from a one sample t-test using SAS (Statistical Analysis System) UNIVARIATE on change from baseline

5. Secondary Outcome: Total Score of Composite Functional Outcomes of Sleep Questionnaire (FOSQ) : Active Phase
Description: The FOSQ was 30-item, validated psychometric instrument that assessed the impact of disorders of excessive sleepiness on functional outcomes relevant to daily behaviors and quality of life (QoL). The responses to the questionnaire were grouped according to five factors for analysis: 1) Activity Level, 2) Vigilance, 3) Intimacy and Sexual Relationships, 4) General Productivity and 5) Social Outcome. Participant used a scale of 0 to 4 to score each question of FOSQ which then grouped in above factors (where 0= I don't do this activity for other reasons, 1= Yes, extreme difficulty, 2= Yes, moderate difficulty, 3= Yes, a little difficulty, and 4= No difficulty). Total score of composite FOSQ was the sum of scores obtained on all 30 questions of the questionnaire. The possible range for the total score of composite FOSQ was from 0-120. A higher total score of composite FOSQ indicates better QoL of the participant.
Time Frame: Day 29
Population: Per protocol population included all participants who fully complied with all study procedures and restrictions. Here, "N" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Participants (Active Phase)
Number analyzed (Participants) | 61
Score on a scale | 17.55 (2.129)

6. Secondary Outcome: Global Self Assessment Score : Active Phase
Description: On Day 29, prior to sleep, participants were asked to rate their overall experience with the strip as compared to before they enrolled in the study: ease of breathing, staying asleep, falling back to sleep, waking up too early, number of awakenings, falling asleep, sleep quality, sleep depth, dry mouth upon awakening, morning headache, nocturia (waking up to urinate), feeling refreshed in the morning. Experience was rated on scale of -2 to 2 were: -2 = Much worse, -1 = Somewhat worse, 0 = No change, 1 = Somewhat improve, 2 = Much improved (higher score indicated improvement).
Time Frame: Day 29
Population: Per protocol population included all participants who fully complied with all study procedures and restrictions. Here, number analyzed signifies participants who were evaluable for the specified categories.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Participants (Active Phase)
Number analyzed (Participants) | 70
Score on a scale
  Ease of breathing: number analyzed (Participants) | 61
  Ease of breathing | 1.4 (0.68)
  Falling asleep: number analyzed (Participants) | 61
  Falling asleep | 0.6 (0.78)
  Staying asleep: number analyzed (Participants) | 61
  Staying asleep | 0.8 (0.76)
  Number of awakenings: number analyzed (Participants) | 61
  Number of awakenings | 0.7 (0.77)
  Falling back to sleep: number analyzed (Participants) | 61
  Falling back to sleep | 0.7 (0.76)
  Waking up too early: number analyzed (Participants) | 61
  Waking up too early | 0.3 (0.63)
  Sleep depth: number analyzed (Participants) | 61
  Sleep depth | 0.7 (0.70)
  Sleep quality: number analyzed (Participants) | 61
  Sleep quality | 0.9 (0.69)
  Nocturia (waking up to urinate): number analyzed (Participants) | 61
  Nocturia (waking up to urinate) | 0.3 (0.60)
  Dry mouth upon awakening: number analyzed (Participants) | 61
  Dry mouth upon awakening | 0.6 (0.82)
  Morning headache: number analyzed (Participants) | 61
  Morning headache | 0.4 (0.67)
  Feeling refreshed in the morning: number analyzed (Participants) | 61
  Feeling refreshed in the morning | 0.8 (0.76)

7. Secondary Outcome: Total Epworth Sleepiness Scale Score (ESS) : Active Phase
Description: Participants answered the following question How likely are you to doze off or fall asleep in the following situations, in contrast to feeling just tired? 1. Sitting and reading, 2. Watching TV, 3. Sitting, inactive in a public place (e.g. a theatre or a meeting), 4. As a passenger in a car for an hour without a break, 5. Lying down to rest in the afternoon when circumstances permit, 6. Sitting and talking to someone, 7. Sitting quietly after a lunch without alcohol, and 8. In a car, while stopped for a few minutes in the traffic. Use the following scale to choose the most appropriate number for each situation: 0 = would never doze, 1 = slight chance of dozing, 2 = moderate chance of dozing, and 3 = high chance of dozing. Total ESS was calculated as the sum of all the individual scores observed for the above mentioned situations. The possible range for total ESS was 0-24. A lower total ESS indicates better sleep.
Time Frame: Day 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | All Participants (Active Phase)
Number analyzed (Participants) | 61
Score on scale | 7.410 (4.6021)

8. Secondary Outcome: Number of Snores Per Hour : Baseline, Active and Nasal Resistance Phase
Description: The Investigator or designee recorded the number of snores per hour during the participant's domiciled sleep visits. Numbers of snores were recorded for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: Per protocol population included all participants who fully complied with all study procedures and restrictions. Here, number analyzed signifies participants who were evaluable at specified timepoints
Measure: Mean (Standard Deviation); unit: Number of snores per hour
Arm/Group | All Participants
Number analyzed (Participants) | 70
Number of snores per hour
  Day 1: number analyzed (Participants) | 69
  Day 1 | 308.18 (216.829)
  Day 8: number analyzed (Participants) | 65
  Day 8 | 299.58 (204.598)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 330.30 (233.635)
  Without strip (Day 30 and 31): number analyzed (Participants) | 48
  Without strip (Day 30 and 31) | 317.76 (208.098)
  With strip (Day 30 and 31): number analyzed (Participants) | 50
  With strip (Day 30 and 31) | 324.92 (190.559)

9. Secondary Outcome: Snoring Percent of Sleep Time : Baseline, Active and Nasal Resistance Phase
Description: The Investigator or designee recorded the snoring percent (%) present in sleep time during the participant's domiciled sleep visits. Snoring % was measured for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of sleep time
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of sleep time
  Day 1: number analyzed (Participants) | 69
  Day 1 | 40.33 (27.444)
  Day 8: number analyzed (Participants) | 65
  Day 8 | 38.70 (25.826)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 42.41 (28.974)
  Without strip (Day 30 and 31): number analyzed (Participants) | 48
  Without strip (Day 30 and 31) | 42.11 (27.167)
  With strip (Day 30 and 31): number analyzed (Participants) | 50
  With strip (Day 30 and 31) | 43.22 (24.704)

10. Secondary Outcome: Average Snore Sound Intensity : Baseline, Active and Nasal Resistance Phase
Description: The Investigator or designee recorded the average snore sound intensity during the participant's domiciled sleep visits. Average snore sound intensity was measured for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Decibels
Arm/Group | All Participants
Number analyzed (Participants) | 70
Decibels
  Day 1: number analyzed (Participants) | 69
  Day 1 | 40.67 (6.278)
  Day 8: number analyzed (Participants) | 65
  Day 8 | 41.85 (6.365)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 44.14 (6.730)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 43.10 (4.780)
  With strip (Day 30 and 31): number analyzed (Participants) | 52
  With strip (Day 30 and 31) | 43.89 (4.628)

11. Secondary Outcome: Peak Sore Sound Intensity : Baseline, Active and Nasal Resistance Phase
Description: The Investigator or designee recorded the peak snore sound intensity during the participant's domiciled sleep visits. Peak snore sound intensity was recorded for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Decibels
Groups:
- All Participants: This was a baseline-controlled study and consisted of 3 phases: baseline phase, 28 days active phase followed by a two-night cross-over nasal resistance phase. In the baseline phase all the participants were applied nasal dilator strip during the sleep laboratory night on Day 1 (Night 1). During the active phase all the participants wore nasal dilator strip over a 1 month in-home use period and returned for sleep laboratory nights after 7 (Day 8, Night 8) and 28 days (Day 29, Night 29) of treatment. The nasal resistance phase consisted of 2 sleep laboratory nights (Day 30 Night 30 and Day 31 Night 31), where the participants were randomized to receive a sequence of either 'strip'/' no strip' or 'no strip'/'strip' as per the randomization schedule
Arm/Group | All Participants
Number analyzed (Participants) | 70
Decibels
  Day 1: number analyzed (Participants) | 69
  Day 1 | 67.84 (9.944)
  Day 8: number analyzed (Participants) | 65
  Day 8 | 66.44 (8.854)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 69.87 (8.876)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 69.48 (13.525)
  With strip (Day 30 and 31): number analyzed (Participants) | 52
  With strip (Day 30 and 31) | 70.28 (11.917)

12. Secondary Outcome: Percentage of Participants With Nasal Breathing Route : Baseline, Active and Nasal Resistance Phase
Description: The Investigator or designee recorded the Nasal breathing route during the participant's domiciled sleep visits. Nasal breathing route was observed for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of participants
  Day 1: number analyzed (Participants) | 69
  Day 1 | 26.38 (27.322)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 27.78 (28.200)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 31.25 (29.558)
  Without strip (Day 30 and 31): number analyzed (Participants) | 48
  Without strip (Day 30 and 31) | 44.71 (31.139)
  With strip (Day 30 and 31): number analyzed (Participants) | 50
  With strip (Day 30 and 31) | 48.40 (28.899)

13. Secondary Outcome: Percentage of Participants With Oro-nasal Breathing Route : Baseline, Active and Nasal Resistance Phase
Description: The Investigator or designee recorded the oro-nasal breathing route during the participant's domiciled sleep visits. Oro-nasal breathing route was observed for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of participants
  Day 1: number analyzed (Participants) | 69
  Day 1 | 70.92 (29.496)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 70.26 (28.578)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 64.44 (32.627)
  Without strip (Day 30 and 31): number analyzed (Participants) | 48
  Without strip (Day 30 and 31) | 51.04 (29.894)
  With strip (Day 30 and 31): number analyzed (Participants) | 50
  With strip (Day 30 and 31) | 47.60 (28.508)

14. Secondary Outcome: Total Sleep Time (TST) : Baseline, Active and Nasal Resistance Phase
Description: TST was measured by overnight polysomnography (PSG) using a computerized system. TST was measured for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | All Participants
Number analyzed (Participants) | 70
Minutes
  Day 1 | 369.54 (52.629)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 371.97 (58.359)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 366.26 (69.722)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 317.98 (91.910)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 304.65 (101.447)

15. Secondary Outcome: Sleep Efficiency (SE) : Baseline, Active and Nasal Resistance Phase
Description: Sleep efficiency [SE, a polysomnography (PSG)] was measured as the percentage of total time in bed spent in sleep. It was calculated as the sum of Stage N1, Stage N2, Stage N3, and REM sleep, divided by the total time in bed and multiplied by 100. SE gives an overall sense of how well the participant slept and was measured for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of sleep time
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of sleep time
  Day 1 | 80.50 (10.631)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 81.66 (10.184)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 82.25 (11.607)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 75.56 (16.095)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 73.63 (19.130)

16. Secondary Outcome: Sleep Onset Latency (SOL) : Baseline, Active and Nasal Resistance Phase
Description: Sleep onset latency (SOL, a PSG parameter) was measured as the duration from the time when lights were turned off (as the participants attempted to sleep) till the time participant fell asleep. Determination of sleep and awake state was based on Electroencephalography (EEG) and behavioral parameters change. SOL was measured for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | All Participants
Number analyzed (Participants) | 70
Minutes
  Day 1 | 13.86 (18.469)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 14.92 (17.275)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 9.69 (8.877)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 14.29 (19.943)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 18.45 (23.937)

17. Secondary Outcome: Arousal Index (AI) : Baseline, Active and Nasal Resistance Phase
Description: Arousal index (AI) is the number of arousals and awakenings, reported as a total number per hour of sleep. AI was measured for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Number of arousals per hour
Arm/Group | All Participants
Number analyzed (Participants) | 70
Number of arousals per hour
  Day 1 | 25.12 (11.308)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 25.24 (10.979)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 25.97 (12.916)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 35.33 (17.250)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 38.33 (20.908)

18. Secondary Outcome: Sleep Architecture (Non-Rapid Eye Movement- Stages N1, N2 and N3) : Baseline, Active and Nasal Resistance Phase
Description: Non-Rapid eye movement (NREM) sleep stage consist of 3 progressively deeper stages of sleep: N1 (transition period from being awake to falling asleep), N2 (where breathing and heart rate began to slow) and N3 (slow wave sleep where body heals and repair itself). Sleep architecture (SA) was measured by the percentage of sleep time spent by the participants in each stage (time spent in each stage to total time spent in NREM, multiplied by 100). SA was measured for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of sleep time
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of sleep time
  % N1: Day 1 | 8.30 (4.123)
  % N1: Day 8: number analyzed (Participants) | 66
  % N1: Day 8 | 7.58 (4.140)
  % N1: Day 29: number analyzed (Participants) | 61
  % N1: Day 29 | 8.46 (5.468)
  % N1: Without strip (Day 29 and 30): number analyzed (Participants) | 51
  % N1: Without strip (Day 29 and 30) | 7.65 (6.896)
  % N1: With strip (Day 29 and 30): number analyzed (Participants) | 51
  % N1: With strip (Day 29 and 30) | 8.82 (11.567)
  % N2: Day 1 | 47.93 (6.881)
  % N2: Day 8: number analyzed (Participants) | 66
  % N2: Day 8 | 48.00 (7.876)
  % N2: Day 29: number analyzed (Participants) | 61
  % N2: Day 29 | 47.12 (6.558)
  % N2: Without strip (Day 29 and 30): number analyzed (Participants) | 51
  % N2: Without strip (Day 29 and 30) | 55.41 (8.129)
  % N2: With strip (Day 29 and 30): number analyzed (Participants) | 51
  % N2: With strip (Day 29 and 30) | 54.71 (10.212)
  % N3: Day 1 | 22.83 (7.249)
  % N3: Day 8 | 22.14 (7.060)
  % N3 at Day 29 | 22.38 (6.779)
  % N3: Without strip (Day 29 and 30): number analyzed (Participants) | 51
  % N3: Without strip (Day 29 and 30) | 19.02 (8.255)
  % N3: With strip (Day 29 and 30): number analyzed (Participants) | 51
  % N3: With strip (Day 29 and 30) | 18.37 (9.654)

19. Secondary Outcome: Total Non-rapid Eye Movement (NREM) and Rapid Eye Movement (REM) Sleep : Baseline, Active and Nasal Resistance Phase
Description: Total NREM (N1, 2, and 3) and REM sleep were calculated as the time spent by a participant in the NREM (measured during stable sleep) and REM sleep stages. Total NREM and REM sleep was measured by overnight PSG using a computerized system for all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | All Participants
Number analyzed (Participants) | 70
Minutes
  NREM: Day 1 | 296.30 (41.046)
  NREM: Day 8: number analyzed (Participants) | 66
  NREM: Day 8 | 294.17 (46.660)
  NREM: Day 29: number analyzed (Participants) | 61
  NREM: Day 29 | 289.48 (52.366)
  NREM: Without strip (Day 30 and 31): number analyzed (Participants) | 51
  NREM: Without strip (Day 30 and 31) | 264.82 (79.545)
  NREM: With strip (Day 30 and 31): number analyzed (Participants) | 51
  NREM: With strip (Day 30 and 31) | 249.63 (81.397)
  REM: Day 1 | 73.10 (20.976)
  REM: Day 8: number analyzed (Participants) | 66
  REM: Day 8 | 77.52 (22.313)
  REM: Day 29: number analyzed (Participants) | 61
  REM: Day 29 | 76.53 (25.039)
  REM: Without strip (Day 30 and 31): number analyzed (Participants) | 51
  REM: Without strip (Day 30 and 31) | 52.84 (23.452)
  REM: With strip (Day 30 and 31): number analyzed (Participants) | 51
  REM: With strip (Day 30 and 31) | 55.04 (28.592)

20. Secondary Outcome: Respiratory Effort Related Arousals (RERA) : Baseline, Active and Nasal Resistance Phase
Description: Respiratory Effort Related Arousal (RERA) was flattening of an inspiratory portion of nasal pressure with increased respiratory effort leading to arousal. The total number of arousals per hour were calculated as RERA. RERA was measured all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: RERA per hour
Arm/Group | All Participants
Number analyzed (Participants) | 70
RERA per hour
  Day 1 | 14.62 (9.006)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 16.80 (9.611)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 16.30 (10.602)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 20.65 (11.789)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 23.88 (13.757)

21. Secondary Outcome: Percentage of Lowest Arterial Oxygen Saturation (SAO2) During Rapid Eye Movement (REM) and Non-rapid Eye Movement (REM) Sleep Stage : Baseline, Active and Nasal Resistance Phase
Description: Arterial oxygen saturation (SAO2) is the fraction of [oxygen]-saturated hemoglobin relative to total hemoglobin (unsaturated + saturated) in the blood. SAO2 in NREM and REM sleep was measured overnight by pulse oximetry with a finger probe using a computerized system. Lowest SAO2 values observed during the NREM and REM sleep were recorded for this endpoint. Oximetry measurements were performed in all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of SAO2
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of SAO2
  REM: Day 1: number analyzed (Participants) | 69
  REM: Day 1 | 91.33 (3.433)
  REM: Day 8: number analyzed (Participants) | 66
  REM: Day 8 | 91.17 (3.476)
  REM: Day 29: number analyzed (Participants) | 61
  REM: Day 29 | 91.34 (3.219)
  REM: Without strip (Day 29 and 30): number analyzed (Participants) | 50
  REM: Without strip (Day 29 and 30) | 92.30 (3.541)
  REM: With strip (Day 29 and 30): number analyzed (Participants) | 48
  REM: With strip (Day 29 and 30) | 92.42 (3.494)
  NREM: Day 1: number analyzed (Participants) | 69
  NREM: Day 1 | 91.01 (3.012)
  NREM: Day 8: number analyzed (Participants) | 66
  NREM: Day 8 | 90.24 (3.684)
  NREM: Day 29: number analyzed (Participants) | 61
  NREM: Day 29 | 90.75 (3.139)
  NREM: Without strip (Day 29 and 30): number analyzed (Participants) | 51
  NREM: Without strip (Day 29 and 30) | 91.88 (3.386)
  NREM: With strip (Day 29 and 30): number analyzed (Participants) | 51
  NREM: With strip (Day 29 and 30) | 91.96 (3.200)

22. Secondary Outcome: Mean Arterial Oxygen Saturation (SAO2) During Sleep Time : Baseline, Active and Nasal Resistance Phase
Description: SAO2 in sleep time was measured overnight by pulse oximetry with a finger probe using a computerized system. Mean of the observed SAO2 values during entire sleep time was reported for this endpoint. Oximetry measurements were performed in all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of SAO2
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of SAO2
  Day 1: number analyzed (Participants) | 69
  Day 1 | 95.70 (1.468)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 95.70 (1.598)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 95.64 (1.528)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 96.69 (1.364)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 96.71 (1.188)

23. Secondary Outcome: Average Oxygen Desaturation During Sleep : Baseline, Active and Nasal Resistance Phase
Description: Oxygen desaturation is the drop in blood's oxygen level per hours of sleep. Average drop in oxygen level during total sleep was measured overnight by pulse oximetry with a finger probe using a computerized system. Oximetry measurements were performed in all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of oxygen desaturation
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of oxygen desaturation
  Day 1: number analyzed (Participants) | 69
  Day 1 | 4.41 (10.980)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 4.68 (11.679)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 3.49 (1.588)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 2.90 (2.385)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 3.33 (2.113)

24. Secondary Outcome: Percentage of Sleep Time With Arterial Oxygen Saturation (SAO2) Greater Than 90% : Baseline, Active and Nasal Resistance Phase
Description: Percent sleep time with SAO2 greater than 90% was measured overnight by pulse oximetry with a finger probe. Oximetry measurements were performed in all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of sleep time
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of sleep time
  Day 1: number analyzed (Participants) | 69
  Day 1 | 98.59 (3.397)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 97.38 (7.383)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 98.21 (4.021)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 98.41 (4.016)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 99.18 (1.381)

25. Secondary Outcome: Percentage of Sleep Time With Arterial Oxygen Saturation (SAO2) Less Than 90% : Baseline, Active and Nasal Resistance Phase
Description: Percent sleep time with SAO2 less than 90% was measured overnight by pulse oximetry with a finger probe. Oximetry measurements were performed in all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of sleep time
Arm/Group | All Participants
Number analyzed (Participants) | 70
Percentage of sleep time
  Day 1: number analyzed (Participants) | 69
  Day 1 | 0.66 (2.863)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 1.29 (6.713)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 0.56 (2.742)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 0.49 (2.533)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 0.12 (0.475)

26. Secondary Outcome: Apnea/Hypopnea Index (AHI) : Baseline, Active and Nasal Resistance Phase
Description: Apnea/Hypopnea Index (AHI) was measured as the number of events (apnea and hypopnea) per hour of sleep. AHI was measured using overnight by PSG using a computerized system. PSG was performed in all participants with strip on Day 1 (Visit 2) in baseline phase, Day 8 (Visit 3) and Day 29 (Visit 4) in active phase, and in participants with and without strip on Day 30 (Visit 5) and Day 31 (Visit 6) cumulatively, in nasal resistance phase.
Time Frame: Day 1, Day 8, Day 29, Day 30 and Day 31
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: AHI events per hour
Arm/Group | All Participants
Number analyzed (Participants) | 70
AHI events per hour
  Day 1 | 4.08 (5.499)
  Day 8: number analyzed (Participants) | 66
  Day 8 | 4.26 (5.273)
  Day 29: number analyzed (Participants) | 61
  Day 29 | 5.07 (7.371)
  Without strip (Day 30 and 31): number analyzed (Participants) | 51
  Without strip (Day 30 and 31) | 6.57 (10.489)
  With strip (Day 30 and 31): number analyzed (Participants) | 51
  With strip (Day 30 and 31) | 7.11 (12.948)

ADVERSE EVENTS:
Time Frame: Upto 31 days
Description: Safety population included all participants to whom the study treatment was dispensed were considered evaluable for the safety population.
Groups:
- Participants With Strip (Nasal Resisatnce Phase): The participants were randomized to receive a sequence of either 'strip'/' no strip' or 'no strip'/'strip' on 2 sleep laboratory nights (Day 30 and Day 31) based on the randomization schedule. This arm represents the participants who applied the strip.
- Participants Without Strip (Nasal Resisatnce Phase): The participants were randomized to receive a sequence of either 'strip'/' no strip' or 'no strip'/'strip' on 2 sleep laboratory nights (Day 30 and Day 31) based on the randomization schedule. This arm represents the participants who did not applied the strip.
Arm/Group | All Participants (Baseline Phase) | All Participants (Active Phase) | Participants With Strip (Nasal Resisatnce Phase) | Participants Without Strip (Nasal Resisatnce Phase)
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/70 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/91 | 1/70 | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/91 | 28/70 | 2/55 | 1/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Baseline Phase) (N=91) | All Participants (Active Phase) (N=70) | Participants With Strip (Nasal Resisatnce Phase) (N=55) | Participants Without Strip (Nasal Resisatnce Phase) (N=55)
Bell's Palsy (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Baseline Phase) (N=91) | All Participants (Active Phase) (N=70) | Participants With Strip (Nasal Resisatnce Phase) (N=55) | Participants Without Strip (Nasal Resisatnce Phase) (N=55)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 2 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 0 | 0
SUNBURN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 4 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 9 | 0 | 0
CLAUSTROPHOBIA (Psychiatric disorders) | 0 | 0 | 1 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 1 | 0 | 0
RHINALGIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
APPLICATION SITE REACTION (General disorders) | 0 | 1 | 0 | 0
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
VIIth NERVE PARALYSIS (Nervous system disorders) | 0 | 1 | 0 | 0
APPLICATION SITE FISSURE (General disorders) | 0 | 1 | 0 | 0
Application site haematoma (General disorders) | 0 | 1 | 0 | 0
BLOOD CHOLESTEROL Increased (Investigations) | 0 | 1 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 1
TINEA PEDIS (Infections and infestations) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.